CLINICAL TRIAL: NCT04996459
Title: Real-world Study of Tislelizumab in the Systematic Treatment of Advanced Hepatocellular Carcinoma
Brief Title: Tislelizumab in the Systematic Treatment of Advanced Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lu Wang, MD, PhD, Head of liver surgery department, Fudan University
Other Study IDs: GWK-2020-06
Record Dates: First submitted 2021-08-04; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tislelizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tislelizumab group
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab 200mg iv q3w

SUMMARY:
Study purpose: To evaluate the efficacy and safety of Tislelizumab in combination with advanced hepatocellular carcinoma in the real world; Study design: Non-intervention, single center, case registration, real-world study; Number of registrations: 40;

Source of data: This project is a non-interventionary real world case follow-up registration. All registration data are from real clinical practice cases. The collected data include the following requirements:

1. Age ≥18 years old;
2. Unresectable hepatocellular carcinoma confirmed by histological examination or clinical diagnosis;
3. Plan or have received systemic therapy combined with Tiralizumab;
4. No participation in other clinical studies;
5. Access to Tislelizumab treatment and other clinical records; Primary endpoint: Overall response rate; Secondary endpoint: Disease control rate, progress free survival, overall survival, safety; Exploratory endpoint: To explore the predictive value of multiple Biomarker combinations, such as PD-L1, TMB, MSI, DDR, POLE/POLD, in HCC immunotherapy response.

ELIGIBILITY:
This project is a non-interventionary real world case follow-up registration. All registration data are from real clinical practice cases. The collected data include the following requirements:

1. Age ≥18 years old;
2. Unresectable hepatocellular carcinoma confirmed by histological examination or clinical diagnosis;
3. Plan or have received systemic therapy combined with Tislelizumab;
4. No participation in other clinical studies;
5. Access to Tislelizumab treatment and other clinical records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients registrated and treated with Tislelizumab at least once were included in the efficacy analysis population as well as the safety analysis population.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
overall response rate | 6 weeks
  overall response rate

SECONDARY OUTCOMES:
disease control rate | 6 weeks
  disease control rate
progress free survival | 6 weeks
  progress free survival
overall survival | 6 weeks
  overall survival
Safety (the incidence of adverse events and serious adverse events) | 3 weeks
  the incidence of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Lu Wang, M.D., Principal Investigator — FUSCC
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China